CLINICAL TRIAL: NCT02136966
Title: Joint Infant and Young Child Nutrition Program in Burkina Faso : Impact Evaluation
Brief Title: Joint Infant and Young Child Nutrition Program and Malnutrition Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: Micronutrient Initiative (Other); Institute of Tropical Medicine, Belgium (Other); Terre des Hommes (Unknown)
Responsible Party: Principal Investigator, Hermann Lanou, Dr, Institut de Recherche en Sciences de la Sante, Burkina Faso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRSS0002
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Growth Failure; Good Infant and Young Child Feeding Practices
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Programme (Experimental): * Distribution of Micronutrients powders (MNP)
  * Intensive counseling on Infant and Young Child Nutrition
  * Cooking demonstrations
  Interventions: Other: MNP + IYCN counseling + cooking demonstrations
- Controle (No Intervention): * Usual Infant growth monitoring and promotion activities
  * No distribution of micronutrients powders
  * No Intensive counseling
  * No cooking demonstrations

INTERVENTIONS:
Other: MNP + IYCN counseling + cooking demonstrations — Growth monitoring and promotion sessions will take place every month at village level for all children 0-23 months of age and will serve as an entry point for all the interventions. During these sessions children under 24 months will be weighed monthly and screened for MAM and uncomplicated SAM for treatment in the community as well as complicated SAM for referral to health facility During the monthly sessions cooking demonstrations will take place in which the community Health workers will instruct the mother how to prepare a good complementary food for 6-23 months olds adding the MNP. These meals will be given to the child during the session. Mothers will be encouraged to prepare the same meal at home During the monthly sessions enhanced IYCN counseling will be given to the mothers of 6-23 months olds, using improved BCI messages developed based on the rapid assessment of practices and foods available in the community and adaptation of the WHO manual.
  Arms: Programme

SUMMARY:
Study title: Joint Infant and young children nutrition program in Burkina Faso: Impact evaluation Hypothesis: The fortification of complementary foods associated with a counseling on feeding practices for infants and young children prevents malnutrition in 6-23 months-old children.

Objective: to assess the effectiveness of a promotional care package in preventing malnutrition among children aged 6-23 months.

DETAILED DESCRIPTION:
The 'Institut de Recherche en Sciences de la Santé (IRSS)', in collaboration with Micronutrient Initiative (MI), the Institute of Tropical Medicine (ITM) Antwerp (Belgium), and the Health District of Tougan, will conduct a study to assess the effectiveness of a promotional package in the prevention and management of malnutrition among children aged 6-23 months.

This promotional package includes:

1. A monthly follow-up sessions promoting growth in which detailed advice on feeding practices infant and young child feeding (IYCF) will be given to the mothers of children 6-23 months . These behavioral change informations be developed based on the rapid assessment of practices and foods available in the community and adaptation of the WHO manual.
2. The distribution of micronutrient powders (MNP) (15 micronutrients) to mothers of children 6-23 months of age for home fortification of complementary foods
3. Intensive counseling sessions and cooking demonstrations every two weeks for moderately malnourished children . Cooking demonstrations will include instructions on adding micronutrient powders and oil to meals .

ELIGIBILITY:
Inclusion Criteria:

* Mothers of 6 to 23 months old children
* Reside in the study area
* Accept to use MNP

Exclusion Criteria:

* Mothers of children aged less than 6 months or more than 23 months.
* Refusal

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2212 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of children with Weight-for-height and/or Height-for-age ZScore <-2 | 1 year

SECONDARY OUTCOMES:
Proportion of mothers who can describe at least 3 best practices about IYCN | 3, 6 and 12 months

OTHER OUTCOMES:
Number of children with adverse events as a safety measure of the use of Micronutrient Powder for food fortification at home | 1 year
  The morbidity will be assess every week from baseline until the end of the intervention (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Lanou, MSc, Principal Investigator — Institut de Recherche en Sciences de la Santé (IRSS), Ouagadougou, Burkina Faso
Locations (1):
- LANOU Hermann Bienou, Ouagadougou, Kadiogo, Burkina Faso

REFERENCES:
- [Derived] Lanou HB, Osendarp SJM, Argaw A, De Polnay K, Ouedraogo C, Kouanda S, Kolsteren P. Micronutrient powder supplements combined with nutrition education marginally improve growth amongst children aged 6-23 months in rural Burkina Faso: A cluster randomized controlled trial. Matern Child Nutr. 2019 Oct;15(4):e12820. doi: 10.1111/mcn.12820. Epub 2019 Jun 10. PMID 30941887